CLINICAL TRIAL: NCT06395870
Title: A Phase I, Open-label Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of LUCAR-G39D, a Dual-targeted Cell Preparation Targeting CD19/CD20, in Patients With Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
Brief Title: Targeting CD19/CD20 Dual-targeted Cell in Patients With Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Principal Investigator, Huilai Zhang, Director of lymphoma department, Tianjin Medical University Cancer Institute and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB2303-0001
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-05

CONDITIONS: B-Cell Non-Hodgkin Lymphoma-Recurrent; B-Cell Non-Hodgkin Lymphoma-Refractory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LUCAR-G39D cells product (Experimental): Each subject will be given a single-dose LUCAR-G39D cells infusion at each dose level.
  Interventions: Biological: LUCAR-G39D cells product

INTERVENTIONS:
Biological: LUCAR-G39D cells product — Prior to infusion of the LUCAR-G39D, subjects will receive a conditioning premedication regimen consisting of cyclophosphamide and fludarabine.

SUMMARY:
A phase I, open-label clinical study to evaluate the safety, tolerability, and efficacy of LUCAR-G39D, a dual-targeted cell preparation targeting CD19/CD20, in patients with relapsed/refractory B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
This is an open-label, dose-escalation/dose extension study to assess the safety, tolerability, and efficacy of LUCAR-G39D in the patient ≥ 18 years of age with relapsed or refractory B-cell non-Hodgkin lymphoma. Subjects who meet the eligibility criteria will receive a single dose of LUCAR-G39D injection. The study will include the following sequential phases: screening, pre-treatment (lymphodepleting chemotherapy), treatment, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects have fully understood the possible risks and benefits of participating in this study, are willing to follow and able to complete all trial procedures, and have signed informed consent.
2. Aged 18-75 years (inclusive).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Histologically confirmed B-cell non-Hodgkin Lymphoma that expresses at least one of CD19/CD20.
5. At least one evaluable tumor lesion according to Lugano 2014 criteria.

Response to prior therapy is consistent with one of the following:

1. Primary refractory.
2. Relapsed or refractory after 2 or more lines of therapy.
3. For LBCL, 3B FL. t-iNHL:

   * Relapse within 12 months after first-line chemoimmunotherapy to achieve CR;
   * Progression or relapse within 12 months after autologous hematopoietic stem cell transplantation;

     7. Life expectancy≥ 3 months 8. Clinical laboratory values meet screening visit criteria

   Exclusion Criteria:

   Subject eligible for this study must not meet any of the following criteria:

   1. Prior antitumor therapy with insufficient washout period ; 2. Patients who received autologous CAR-T cell therapy (except CD19-targeted) or autologous gene therapy; 3. Patients who received allogeneic hematopoietic stem cell transplantation or allogeneic therapy; 5. Patients who are positive for any index of hepatitis B surface antigen (HBsAg), hepatitis B virus deoxyribonucleic acid (HBV DNA), hepatitis C antibody (HCV-Ab), hepatitis C virus ribonucleic acid (HCV RNA), or human immunodeficiency virus antibody (HIV- Ab).

   6. Known life-threatening allergies, hypersensitivity, or intolerance to LUCAR-G39D CAR-T cell or its excipients, including DMSO.

   7. Pregnant or lactating women;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity and type of TEAEs (Treatment-emergent Adverse Events) | Through study completion , an average of 2 years after LUCAR-G39D infusion (Day 1)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Pharmacokinetics in peripheral blood | Through study completion , an average of 2 years after LUCAR-G39D infusion (Day 1).
  CAR positive T cells and CAR transgene levels in peripheral blood after LUCAR-G39D infusion.
Pharmacokinetics in bone marrow | Through study completion , an average of 2 years after LUCAR-G39D infusion (Day 1)
  CAR positive T cells and CAR transgene levels in bone marrow after LUCAR-G39D infusion.
The recommended Phase II dose (RP2D) for this cell therapy | Within 30 days after LUCAR-G39D infusion
  RP2D established through ATD+BOIN design and the DLTs occurring following CAR T-cell infusion.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Through study completion, an average of 2 years after LUCAR-G39D infusion (Day 1)
  Objective Response Rate (ORR) is defined as the proportion of subjects who achieve CR or PR after treatment via LUCAR-G39D cell infusion
Progression-free survival (PFS) | Through study completion, an average of 2 years after LUCAR-G39D infusion (Day 1)
  Progression Free Survival (PFS) is defined as the time from the date of first infusion of the LUCAR-G39D to the first documented disease progression (according to Lugano 2014) or death (due to any cause), whichever occurs first
Overall Survival (OS) | Through study completion, an average of 2 years after LUCAR-G39D infusion (Day 1)
  Overall Survival (OS) is defined as the time from the date of first infusion of LUCAR-G39D to death of the subject
Time to Response (TTR) | Through study completion, an average of 2 years after LUCAR-G39D infusion (Day 1)
  Time to Response (TTR) is defined as the time from the date of first infusion of LUCAR-G39D to the date of the first response evaluation of the subject who has met all criteria for CR or PR.
Duration of Response (DoR) | Through study completion, an average of 2 years after LUCAR-G39D infusion (Day 1)
  Duration of Remission (DoR) is defined as the time from the first documentation of remission (CR or PR) to the first documented relapse evidence of the responders.
Immunogenicity assessment of LUCAR-G39D cells | Through study completion, an average of 2 years after LUCAR-G39D infusion (Day 1)
  The incidence of Anti- LUCAR-G39D antibody in patients who received LUCAR-G39D cells infusion

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Oncology Department, The First Affiliated Hospital of USTC west district, Hefei, Anhui
  - Tianjin Cancer Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No